CLINICAL TRIAL: NCT07142538
Title: The Effect of an 8-Week Corrective Exercise Programme on the Tone and Viscoelastic Properties of Back Muscles in Thoracic Kyphosis
Brief Title: the Tone and Viscoelastic Properties of Back Muscles in Thoracic Kyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, director, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hakanpolat3
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Exercise; Kyphosis
MeSH Terms: conditions — Motor Activity; Kyphosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corrective exercise group (Active Comparator): 8 weeks, 3 days a week, 45 minutes shoulder, neck and back exercises postur exercises
  Interventions: Other: exercises
- control group (Active Comparator): Shoulder and neck posture exercises Home exercises 8 weeks 3 days a week
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Exercise training was provided to both groups.

SUMMARY:
The thoracic curvature of the spinal column occurs in the sagittal plane. While the normal thoracic kyphosis angle of the spine is 20-40°, an angle of 45-50° is referred to as postural kyphosis, increased kyphosis, or hyperkyphosis. The strength of the central and deep back muscles of the trunk controls spinal stability and intervertebral movements in dynamic situations. This ensures that thoracic curvature is maintained within normal physiological limits.

Increased kyphosis can result from poor postural habits, prolonged computer use, trunk asymmetry, and muscle weakness. Studies have reported an increase in thoracic kyphosis, postural deviations in the trunk, and changes in shoulder and head positions as a result of weakening of the back muscles. Corrective exercise programmes aimed at strengthening the back muscles are frequently used in the treatment of thoracic kyphosis. The effects of exercise programmes on muscle strength, endurance, and kyphosis angle have been investigated. However, there are few studies examining the effects of corrective exercise programmes on muscle tone and viscoelastic properties in the back muscles. In our study, we aim to investigate the effects of an 8-week corrective exercise programme on the tone and viscoelastic properties of the back muscles in individuals with thoracic kyphosis and to propose its inclusion as a contemporary approach in clinical treatment protocols.

DETAILED DESCRIPTION:
The thoracic curvature of the spinal column occurs in the sagittal plane. While the normal thoracic kyphosis angle of the spine is 20-40°, an angle of 45-50° is referred to as postural kyphosis, increased kyphosis, or hyperkyphosis. The strength of the central and deep back muscles of the trunk controls spinal stability and intervertebral movements in dynamic situations. This ensures that thoracic curvature is maintained within normal physiological limits.

Increased kyphosis can result from poor postural habits, prolonged computer use, trunk asymmetry, and muscle weakness. Studies have reported an increase in thoracic kyphosis, postural deviations in the trunk, and changes in shoulder and head positions as a result of weakening of the back muscles. Corrective exercise programmes aimed at strengthening the back muscles are frequently used in the treatment of thoracic kyphosis. The effects of exercise programmes on muscle strength, endurance, and kyphosis angle have been investigated. However, there are few studies examining the effects of corrective exercise programmes on muscle tone and viscoelastic properties in the back muscles. In our study, we aim to investigate the effects of an 8-week corrective exercise programme on the tone and viscoelastic properties of the back muscles in individuals with thoracic kyphosis and to propose its inclusion as a contemporary approach in clinical treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* having a kyphosis degree of ≥50° in individuals with thoracic kyphosis and voluntarily participating in the study.

Exclusion Criteria:

* individuals with scoliosis, Scheuermann's kyphosis, and other congenital spinal problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
The MyotonPro | 8 weeks
  device can determine the stiffness, tone, and elasticity properties of muscles. This previously calibrated device creates a mechanical stimulus that induces the damped natural oscillations of the tissues using a 3 mm diameter probe placed perpendicular to the muscle with a non-invasive handheld feature. The resulting oscillations are recorded by an accelerometer. MyotonPro® is a valid and reliable method for determining muscle tone, stiffness, and elasticity, and it also offers high test-retest reliability and reproducibility .
Flexible Ruler: | 8 weeks
  The flexible ruler method is a reliable method used to measure cervical, thoracic, and lumbar spine curvature. The measurement is taken using a 40 cm long flexible ruler while standing with arms relaxed at the sides, head upright, and eyes looking straight ahead. The C2 and C7 vertebrae are palpated and marked using removable adhesive skin markers. The flexible ruler is then placed over the cervical lordosis between these two points, and markers indicating the location of the C2 and C7 spinous processes are placed on it. The flexible ruler is placed on millimeter paper, and the resulting curve is reflected. A vertical angle is drawn from the peak of the curve to the baseline, and the cervical lordosis deviation angle is determined using an angle-to-angle connection
Kyphosis-Specific Spine Appearance Questionnaire | 8 weeks
  The Kyphosis-Specific Spine Appearance Questionnaire consisted of 10 items on a Likert scale (1 to 5) regarding patients' perceptions of appearance; higher scores indicated worsening deformity and increased concern about kyphosis-specific appearance. The first item is based on drawings showing varying degrees of severity of hyperkyphosis deformity in the sagittal plane. Questions two through ten are based on textual questions that rate concerns about other aspects of spinal deformity appearance. The total score of the questionnaire is calculated as the average of the ten responses

CONTACTS AND LOCATIONS:
Locations (1):
- SANKO University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No